CLINICAL TRIAL: NCT06653413
Title: Exploring the Diagnostic Performance of Dynamic Chest Radiology in Chronic Obstructive Pulmonary Disease
Status: Enrolling by invitation | Type: Observational
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: NFEC-2024-158; 32470763 (Other Grant/Funding Number: Chinese National Natural Science Foundation project)
Record Dates: First submitted 2024-10-20; First posted 2024-10-22 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: Chronic obstructive pulmonary disease; Dynamic chest radiology; Pulmonary function test; Diagnosis
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COPD group: any patient who complains of dyspnea, chronic cough or sputum, a history of recurrent lower respiratory infection and/or a history of exposure to disease risk factors, Pulmonary function examination indicated that FEV1/FVC <0.7 after bronchodilator was used to confirm COPD.
- normal group: No acute or chronic cardiopulmonary disease in the past, no abnormal lung physical examination and lung imaging examination in the past month, no history of infectious diseases.

SUMMARY:
The prevalence of chronic obstructive pulmonary disease (COPD) is on the rise, leading to an increasing economic and social burden. Currently, the diagnosis and staging of COPD heavily rely on pulmonary function testing. However, limitations such as patient cooperation and comorbidities can hinder accurate diagnosis. In situations like a respiratory pandemic, pulmonary function testing may not be feasible. Dynamic chest radiography has emerged as a promising area of research due to its quick procedure, high patient cooperation, low risk, minimal radiation exposure, and reduced direct contact. Recent clinical studies have started to explore the relationship between dynamic chest X-ray measurements and lung function parameters. However, there is a noticeable scarcity of research focusing on the use of dynamic chest X-ray in aiding the diagnosis of COPD, particularly in Chinese populations where cohort data is lacking. Consequently, there is a pressing need to investigate the correlation between various dynamic chest radiograph parameters and lung function indicators, as well as their potential diagnostic value in COPD.

DETAILED DESCRIPTION:
The incidence and mortality of COPD continue to rise in China, but the awareness level of patients with this disease is not enough. Due to the low treatment compliance, it is not possible to conduct regular review, resulting in difficult to effectively control the disease, acute aggravation of repeated attacks, and then bring a heavy economic burden to society. Therefore, in order to reduce the occurrence of acute exacerbations and improve the quality of life of patients, COPD patients need to strengthen their awareness of the disease, improve treatment compliance, and undergo regular review.

The severity of COPD is diagnosed and assessed mainly by pulmonary function examination. Lung capacity, lung volume, and lung diffusion capacity can be determined by a lung function test to assess the health of lung function. Airflow limitation is an important diagnostic criterion, and the key indicator for determining airflow limitation is the one-second rate (FEV1/FVC) less than 0.7 after inhalation of bronchodilators. The percentage of measured forced expiratory volume in the first second to the estimated value (FEV1%pred) was the primary parameter for assessing the severity of COPD. However, some literature has pointed out that FEV1%pred does not fully reflect the clinical symptoms and quality of life of patients. Although pulmonary function examination is of great significance in evaluating patients' lung conditions, it can not fully evaluate small airway lesions and lung parenchymal injury, and there are problems of non-standard and inaccurate data. Due to the low rate of pulmonary function examination, it can not fully represent the lung condition of patients, and it is still necessary to combine other examination methods to comprehensively evaluate the lung health status of patients.

Dynamic Chest Radiography (DCR) is a real-time X-ray imaging system that takes continuous images of a moving chest, usually in 10 to 20 seconds, and is a fast, well-tolerated, and simple chest radiography technique. Measurements of diaphragm movement, lung area, and lung perfusion can provide multiple examination information for COPD patients and supplement baseline deficiencies in critically ill patients.

The purpose of this study was to evaluate the dynamic chest radiography of COPD patients based on Chinese population, analyze the characteristics of dynamic chest radiography of COPD patients, and study the correlation between chest radiography and lung function. To study the value of dynamic chest radiography in diagnosing COPD. To investigate the role of dynamic chest radiography in evaluating the severity of airflow restriction in COPD and predicting the clinical outcome of COPD. Through multidimensional dynamic assessment of patients, dynamic chest radiography can help doctors more accurately diagnose patients' conditions, and timely interventional treatment, so as to reduce the occurrence of acute exacerbations, delay the risk of disease progression, and improve patients' quality of life.

ELIGIBILITY:
Inclusion Criteria:

- COPD group: (1) Patients ≥30 years of age and ≤ 80 years of age who meet the 2023 GOLD Guidelines for the Diagnosis and Treatment of Chronic Obstructive Pulmonary Disease, i.e., anyone who complains of dyspnea, chronic cough or sputum, a history of recurrent lower respiratory infection and/or exposure to disease risk factors, Moreover, pulmonary function examination indicated that FEV1/FVC <0.7 after bronchodilator was used to confirm COPD. FEV1%pred is used to determine the severity of airflow obstruction: Grade GOLD 1 (mild) : FEV1%pred ≥ 80%, Grade GOLD2 (moderate) : 50% ≤ FEV1%pred < 80%, grade GOLD3 (severe) : 30% ≤ FEV1%pred < 50%, GOLD4 grade (extremely severe) : FEV1%pred < 30%; (2) Signing informed consent; (3) Can cooperate with the completion of dynamic chest X-ray (complete dynamic chest X-ray positioning for 20 seconds, during which calm breathing, hard breathing, can hold breath for at least 7 seconds).

Normal Group: (1) Age ≥30 years old and ≤ 80 years old; (2) Normal pulmonary ventilation function; (3) Exclude chronic airway diseases (such as COPD, asthma, bronchiectasis, etc.); (4) Signing informed consent; (5) Can cooperate with the completion of dynamic chest X-ray (complete dynamic chest X-ray positioning for 20 seconds, during which calm breathing, hard breathing, can hold breath for at least 7 seconds).

Exclusion Criteria:

* COPD group: (1) A history of cancer, lung surgery, other lung diseases (such as pneumonia, active tuberculosis, severe bronchiectasis); (2) Combined with muscle-related diseases such as myasthenia gravis or wasting diseases that affect muscle mass such as severe hyperthyroidism and advanced malignant diseases; (3) Pregnant or lactating women; (4) Significant radiation exposure (dose >10mSv) was involved in the 12 months prior to study participation. Normal Group: (1) Have acute or chronic cardiopulmonary disease in the past, abnormal lung physical examination and lung imaging examination in the past, and have a history of infectious diseases within the past 1 month; (2) Pregnant or lactating women; (3) Significant radiation exposure (dose >10mSv) was involved in the 12 months prior to study participation.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This is a prospective clinical study of COPD patients and normal subjects in our hospital. This study has been approved by the hospital Ethics Committee and the patient's informed consent has been obtained (approval number: MR-44-24-016286).
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Dynamic chest radiographs were used to measure diaphragm movement, lung field area and lung field area change rate | 3 year
  Dynamic chest radiographs of patients with COPD were analyzed and their correlation with lung function was studied. To study the value of dynamic chest radiography in diagnosing COPD. To investigate the role of dynamic chest radiography in evaluating the severity of airflow restriction in COPD and predicting the clinical outcome of COPD.

CONTACTS AND LOCATIONS:
Overall Officials: Laiyu Liu, professor, Study Chair — Nanfang Hospital, Southern Medical University
Locations (1):
- Guangdong Locations, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yu D, Xie W, Guo Y, Zhu X, Liang W, Li M, Mao Y, He Z, Wu J, Yuan L, Huang W, Huang J, He S, Zhou Z, Huang X, Zhan Y, Dong H, Cai S, Cui ZK, Qin G, Liu L. Dynamic Chest Radiography as an Alternative to Pulmonary Function Tests for Chronic Obstructive Pulmonary Disease. Radiology. 2025 Dec;317(3):e251296. doi: 10.1148/radiol.251296. PMID 41400467